CLINICAL TRIAL: NCT03311178
Title: An International Multicentre Open-label Comparative Therapeutic Exploratory Trial to Investigate the Role of a New Neonatal Formulation of Dobutamine in the Treatment of Haemodynamic Insufficiency in the Immediate Postnatal Period
Brief Title: Dobutamine in the Treatment of Haemodynamic Insufficiency in the Immediate Postnatal Period
Acronym: NeoCirc-001
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Substudy 001B is not required at this stage of the PIP
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz (Other)
Collaborators: Hospital Universitario La Paz (Other); Brighton and Sussex University Hospitals NHS Trust (Other); University of Luebeck (Other); Servicio Vasco de Salud Osakidetza, Spain (Unknown); University of Liverpool (Other); Vest Children´s Hospital, Germany (Unknown); Datteln University Witten-Herdecke (Unknown); Iuliu Hatieganu University of Medicine and Pharmacy (Other); Semmelweis University (Other); University of Pecs (Other); Gazi University (Other); Tufts Medical Center (Other); Hannover Medical School (Other); Onorach Clinical Dundee, Scotland (Unknown); Proveca Limited Daresbury, England (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Adelina Pellicer, Chief Investigator, Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neocirculation 001
Record Dates: First submitted 2014-05-27; First posted 2017-10-17 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Shock
Keywords: Shock; Preterm infant; Dobutamine
MeSH Terms: conditions — Shock; Premature Birth | interventions — Dobutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dobutamine (Experimental): Infants who meet the definition of poor perfusion state will be treated at the discretion of the responsible physician following the standard local policies. The interventions will be dobutamine from a new neonatal formulation developed for NeoCirc and/or other treatments (including any other cardiovascular drug or volume replacement with normal saline).
  Interventions: Drug: Dobutamine

INTERVENTIONS:
Drug: Dobutamine — Infants who meet the definition of poor perfusion state will be treated at the discretion of the responsible physician following the standard local policies. The interventions will be dobutamine from a new neonatal formulation developed for NeoCirc and/or other treatments (including any other cardiovascular drug or volume replacement with normal saline).

SUMMARY:
Haemodynamic insufficiency after birth is seen commonly in babies born prematurely and is associated with adverse outcomes. In current clinical practice, a combination of blood pressure and clinical signs is used to guide therapy. However, blood pressure is a poor surrogate of systemic and organ (brain) blood flow distribution during transitional circulation. This state is characterised by increased peripheral vascular resistance and increased afterload causing myocardial depression and impaired blood flow distribution in spite of 'normal' blood pressure. Echocardiography-Doppler (Echo-D) measurement of superior vena cava (SVC) flow has been proposed as a more clinically relevant marker of circulatory impairment shortly after birth than systemic hypotension. When there is low SVC flow, several small-scale clinical trials have suggested dobutamine as the optimal therapeutic option. However the associations between SVC flow and short- and long- term outcomes are not strong enough to allow SVC flow alone to be the basis for the inclusion of patients into a confirmatory trial to demonstrate the efficacy and safety of dobutamine.

NeoCirc-001 - The primary objective is to answer some important questions required for the design of a subsequent placebo-controlled trial (NeoCirc-003), which will evaluate the effectiveness of a new neonatal formulation of dobutamine to treat haemodynamic insufficiency in the first 72 hours after birth in babies born at less than 33 weeks' gestation. Observational data will be collected from this population with a view to determining the degree to which diagnostic measures influence treatment decisions. The primary outcome is death or worst cranial ultrasound (CUS) appearance at or before 36 weeks' gestation.

NeoCirc-001A - The primary objective is to estimate the elimination half-life, and consequently the time to steady-state of dobutamine in extremely premature neonates.

NeoCirc-001B - The primary objective is to construct a population pharmacokinetic pharmacodynamic model that will be validated using samples collected during the confirmatory trial (NeoCirc-003).

ELIGIBILITY:
Inclusion criteria for NeoCirc-001, 001A and 001B -

Target population for informed consent:

* neonates 24 to 32+6 weeks´ gestation,
* postnatal age <72 hours;

Infants eligible for circulatory failure pathway:

* parental informed consent obtained;
* The infants will be assessed, as per routine clinical practice, for clinical signs indicating infants at risk of poor perfusion, and will be recruited if they develop haemodynamic insufficiency defined as: either two or more of: (i) Mean blood pressure (MBP) < gestational age (GA)-1 mmHg (invasive/non-invasive, two readings 15 min apart); (ii) SVC flow < 51 ml/kg/min; (iii) capillary refill time (CRT) > 4 sec; (iv) Lactate > 4 mmol/l (v) Base excess <-9 mmol/l or: MBP < GA -5 mmHg (invasive/non-invasive, two readings 15 min apart)

Exclusion Criteria: NeoCirc-001, 001A and 001B -

* non-viability;
* congenital hydrops or malformations likely to affect cardiovascular adaptation;
* surgery planned within 72 hours of birth;
* chromosomal anomalies;
* informed consent form (ICF) not signed.

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2014-05-30 (Actual); Primary Completion 2015-10-13 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Mortality, or intraventricular haemorrhage (IVH) grades 3 or 4, or cystic and non-cystic periventricular leukomalacia (PVL), or porencephalic cysts, ventriculomegaly, or cerebellar haemorrhage. | at 36 (+/-2 weeks) postmenstrual age
  A composite endpoint is defined as follows: treatment failure is when one of the following is true at or before gestational age 36 (+/-2 weeks), when all surviving patients will have a cranial ultrasound (CUS)-
  1. Neonate dies, or
  2. Intraventricular haemorrhage (IVH) grades 3 or 4, or
  3. cystic and non-cystic periventricular leukomalacia (PVL), or
  4. porencephalic cysts, ventriculomegaly, or cerebellar haemorrhage.
Half-life of the neonatal formulation of dobutamine. | The first sample will be drawn after the end of the infusion, at the time when dobutamine ceases. The second sample will be taken at different study time points after the end of infusion (from 5 min to 6 hours).
  NeoCirc-001A: Half-life of the neonatal formulation of dobutamine.
  The first sample will be drawn after the end of the infusion, at the time when dobutamine ceases reaching the systemic circulation of the neonate, defined as time end (te). To calculate the end of infusion (te) the dead space used in each unit will be taken into account (see below). The second sample will be taken at different study time points after the end of infusion:
  * 5 min after te
  * 15 min after te
  * 45 min after te
  * 2 hours after te
  * 6 hours after te Two infants will be allocated to each time point. Sampling times will be assigned randomly to the patients.

SECONDARY OUTCOMES:
Arterial blood pressure | First 72 hours of life (data collection every 9 ±3 hrs)
  Short-term outcomes of biomarkers for circulatory assessment while a patient is receiving cardiovascular support
Capillary refill time | First 72 hours of life (data collection every 9 ±3 hrs)
  Short-term outcomes of biomarkers for circulatory assessment while a patient is receiving cardiovascular support
Urine output | First 72 hours of life (data collection every 9 ±3 hrs)
  Short-term outcomes of biomarkers for circulatory assessment while a patient is receiving cardiovascular support
Blood lactate concentration | First 72 hours of life (data collection every 9 ±3 hrs)
  Short-term outcomes of biomarkers for circulatory assessment while a patient is receiving cardiovascular support
Base excess | First 72 hours of life (data collection every 9 ±3 hrs)
  Short-term outcomes of biomarkers for circulatory assessment while a patient is receiving cardiovascular support
cerebral regional tissue oxygen saturation (rStO2) | First 72 hours of life (data collection every 6 ±1 hrs)
  Cerebral regional tissue oxygen saturation (rStO2) measured by means of near-infrared spectroscopy
Background pattern | First 72 hours of life (data collection every 6 ±1 hrs)
  Background pattern measured by means of Amplitude-integrated electroencephalography (aEEG/EEG)
Superior vena cava flow | First 72 hours of life (data collection every 9 ±3 hrs)
  Short-term outcomes of biomarkers for circulatory assessment while a patient is receiving cardiovascular support
Right cardiac output | First 72 hours of life (data collection every 9 ±3 hrs)
  Short-term outcomes of biomarkers for circulatory assessment while a patient is receiving cardiovascular support
Cerebral fractional oxygen extraction (FOE) | First 72 hours of life (data collection every 6 ±1 hrs)
  FOE= [peripheral oxygen saturation (SaO2)-rStO2] /SaO2
Interburst interval (IBI) | First 72 hours of life (data collection every 6 ±1 hrs)
  Interburst interval (IBI) measured by means of Amplitude-integrated electroencephalography (aEEG/EEG)
Discontinuity | First 72 hours of life (data collection every 6 ±1 hrs)
  Discontinuity measured by means of Amplitude-integrated electroencephalography (aEEG/EEG)
Amplitude | Fist 72 hours of life (data collection every 6 ±1 hrs)
  The amplitude measured by means of aEEG/EEG
Presence of abnormal transients | First 72 hours of life (data collection every 6 ±1 hrs)
  The presence of abnormal transients measured by means of aEEG/EEG
Synchrony | First 72 hours of life (data collection every 6 ±1 hrs)
  The synchrony measured by means of aEEG/EEG
Mortality | From birth to 36 (+/-2 weeks) postmenstrual age
Intraventricular haemorrhage 2-4 | From birth to 36 (+/-2 weeks) postmenstrual age
Survival free of severe brain injury | From birth to 36 (+/-2 weeks) postmenstrual age
  Survival free of severe brain injury measured by means of cranial ultrasound studies
Hypotension | From birth to 36 (+/-2 weeks) postmenstrual age
Hypertension | From birth to 36 (+/-2 weeks) postmenstrual age
Necrotizing enterocolitis | From birth to 36 (+/-2 weeks) postmenstrual age
Patent ductus (PDA) | From birth to 36 (+/-2 weeks) postmenstrual age
Retinopathy of prematurity | at 36 (+/-2 weeks) postmenstrual age
Chronic lung disease | at 36 (+/-2 weeks) postmenstrual age
Oxygen-dependency at discharge | At discharge
early infection | From birth to 72 hours after birth
Nosocomial infection | From birth to 36 (+/-2 weeks) postmenstrual age

OTHER OUTCOMES:
Number of participants with adverse events | Daily during the first four days of life, at 36±2 weeks' gestation or discharge and at 38±2 weeks' gestation or discharge
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Adelina Pellicer, MD PhD, Study Chair — SERMAS La Paz University Hospital; Heike Rabe, MD PhD, Study Director — Brighton and Sussex University Hospitals (BSUH); Fernando Cabañas, MD PhD, Principal Investigator — Servicio Madrileño de Salud (SERMAS)
Locations (1):
- La Paz University Hospital, Department of Neonatology, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kluckow M, Evans N. Low superior vena cava flow and intraventricular haemorrhage in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2000 May;82(3):F188-94. doi: 10.1136/fn.82.3.f188. PMID 10794784
- [Background] Kluckow M, Evans N. Superior vena cava flow in newborn infants: a novel marker of systemic blood flow. Arch Dis Child Fetal Neonatal Ed. 2000 May;82(3):F182-7. doi: 10.1136/fn.82.3.f182. PMID 10794783
- [Background] Osborn DA, Paradisis M, Evans N. The effect of inotropes on morbidity and mortality in preterm infants with low systemic or organ blood flow. Cochrane Database Syst Rev. 2007 Jan 24;2007(1):CD005090. doi: 10.1002/14651858.CD005090.pub2. PMID 17253539
- [Background] Dempsey EM, Barrington KJ. Treating hypotension in the preterm infant: when and with what: a critical and systematic review. J Perinatol. 2007 Aug;27(8):469-78. doi: 10.1038/sj.jp.7211774. PMID 17653217